CLINICAL TRIAL: NCT03342937
Title: A Single Arm, Phase II Study of Pembrolizumab, Oxaliplatin, and Capecitabine in the First Line Treatment of Patients With Gastro-esophageal Cancer.
Brief Title: KeyLargo: Pembrolizumab + Oxaliplatin + Capecitabine in Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00080566
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Results first posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-02

CONDITIONS: Gastric Cancer; Esophagus Cancer
Keywords: pembrolizumab; XELOX; gastric cancer
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oxaliplatin+Capecitabine+Pembrolizumab (Experimental)
  Interventions: Drug: Oxaliplatin+Capecitabine+Pembrolizumab

INTERVENTIONS:
Drug: Oxaliplatin+Capecitabine+Pembrolizumab — For each cycle: Oxaliplatin 130 mg/m2 IV on Day1, Capecitabine 825 or 1000 mg/m2 PO, BID Days on Days1-14, Pembrolizumab 200 mg IV on Day 1.
  This study has 2 parts:
  1. Safety validation part: all Cycles are 21 days in length.
  2. Dose Expansion part: Cycle 1 is 28 days in length. Cycle 2 and beyond are 21 days.

SUMMARY:
This study will be conducted in two stages: 1) safety validation and 2) dose expansion

1. Safety Validation Cohort: The first portion of the study will preliminarily establish the tolerability of the combination of pembrolizumab, oxaliplatin and capecitabine. Five (5) subjects will be enrolled and their safety data after 21 days of treatment will be reviewed before additional subjects are enrolled. Subjects on this portion of the study will only be enrolled at the Duke Cancer Institute.
2. Dose Expansion Cohort: The second portion of the study (ie. phase II) will enroll 30 subjects. In the dose expansion cohort, the first cycle will be modified to allow one week of pembrolizumab monotherapy before starting capecitabine and oxaliplatin (XELOX) chemotherapy, which will allow analysis of biomarkers related to pembrolizumab. Subjects on this portion of the study will be enrolled at the Duke Cancer institute and select external collaborating institutions.

The primary objective of this trial is to describe the progression free survival (PFS) associated with the combination of pembrolizumab, oxaliplatin and capecitabine (pembrolizumab +XELOX) in all patients with previously untreated metastatic esophagogastric adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically documented and radiographically measurable (by RECIST 1.1) adenocarcinoma of the esophagus or stomach (HER2-positive or negative) that is metastatic/recurrent and not amenable to potentially curative treatment
* No prior chemotherapy for metastatic/recurrent disease. Prior adjuvant or neo-adjuvant treatment with a fluoropyrimidine or fluoropyrimidine based regimen is allowed only if it is completed at least 6 months prior to the start of study drug, whether given alone or with radiation therapy. Patients who have received prior neo-adjuvant therapy (chemotherapy and/or radiation therapy) which did not contain 5-FU or capecitabine and have been diagnosed with metastatic disease (with no previous treatment in the metastatic setting) are eligible. No 6-months window is required for these patients. In the setting of metastatic disease requiring local palliation, only radiosensitizing doses of 5-FU or capecitabine monotherapy are permitted.
* Prior radiation therapy is permitted, provided is completed at least 28 days prior to the start of study drug.
* Age ≥ 18 years with ability to understand and willingness to provide informed consent.
* ECOG performance status of 0 or 1.
* Adequate organ and marrow function as defined below by the following:

  1. Absolute neutrophil count (ANC) ≥ 1500 µl
  2. Platelets ≥ 100,000/µl
  3. Hemoglobin (Hgb) ≥ 9 g/dL
  4. Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
  5. AST/ALT ≤ 2 x ULN without liver metastasis; ≤ 5 x ULN with liver metastasis
  6. Creatinine clearance ≥ 50 cc/min

Exclusion Criteria:

* Prior therapy with an anti-PD-1, anti PD-L1, anti-PD-L2, anti-CD137 antibody, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) agents.
* Chemotherapy, targeted small molecule therapy, radiotherapy, experimental agents, prior therapy with anti-tumor vaccines or other immune-stimulatory antitumor agents, or biological cancer therapy (including monoclonal antibodies) within 14 days prior to the start of study drug, or not recovered (≤ grade 1 or baseline) from adverse events due to a previously administered agent.
* Known CNS metastases and/or carcinomatous meningitis. Patients with radiated or resected lesions are permitted, provided the lesions are fully treated and inactive, patients are asymptomatic, and no steroids have been administered for at least 30 days prior to the start of study drug.
* Documented history of clinically significant autoimmune disease (other than well-controlled hypothyroidism) or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo, type I diabetes mellitus, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Receiving systemic steroid therapy or any form of immunosuppressive therapy within 1 week prior to the start of study drug.
* Received a live vaccine within 4 weeks prior to the start of the study drug.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Known history of HIV seropositivity, hepatitis C virus, acute or chronic active hepatitis B infection, or other serious chronic infection requiring ongoing treatment. Patients receiving prophylactic antibiotics (e.g., for prevention of urinary tract infection or chronic obstructive pulmonary disease) are eligible.
* Pregnant or breastfeeding
* Not willing to use an effective method of birth control
* Concurrent severe and/or uncontrolled medical conditions, which may compromise participation in the study, including impaired heart function or clinically significant heart disease.
* Current use of medication specified by the protocol as prohibited for administration in combination with the study drug. This includes patients with a condition requiring systemic treatment with either corticosteroids (>10mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to the start of study drug. Inhaled or topical steroids and adrenal replacement doses > 10mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Recent or current active infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment within 2 weeks prior to the start of study drug.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to the start of study drug (56 days for hepatectomy, open thoracotomy, major neurosurgery) or anticipation of need for major surgical procedure during the course of the study (except fot rhe planned metastatectomy).
* Serious, non-healing wound, ulcer, or bone fracture.
* History of myocardial infarction, NYHA lass III or IV congestive heart failure, arrhythmia requiring therapy, unstable angina, cardia or other vascular stenting, angioplasty, or surgery within 6 months prior to the start of study drug.
* History of other carcinomas within the last five years, except cured non-melanoma skin cancer, curatively treated in-situ cervical cancer, or localized prostate cancer with a current PSA of < 1.0mg/dL on 2 successive evaluations, at least 3 months apart, with the most recent evaluation no more than 4 weeks prior to the start of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hope Uronis, MD, Principal Investigator — Duke University
Locations (7):
- United States (7):
  - Johnston Health Services Corporation, Clayton, North Carolina
  - Duke Cancer Center, Duke University, Durham, North Carolina
  - Maria Parham Healthcare Association, Henderson, North Carolina
  - Scotland Health Care System, Laurinburg, North Carolina
  - Southeastern Regional Medical Center, Lumberton, North Carolina
  - Johnston Health Services Corporation, Smithfield, North Carolina
  - Lexington Medical Center, West Columbia, South Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited at Duke University Medical Center and Lexington Medical Center.
Pre-assignment Details: 36 subjects consented and received the study drugs. 6 subjects received study drugs in the safety run-in. The safety run-in was intended to identify dose-limiting toxicity. No DLTs were observed in the safety run-in and the drug dose levels were not changed in the expansion cohort, therefore; results were for safety validation and expansion were combined.
Groups:
- Oxaliplatin + Capecitabine + Pembrolizumab: For each cycle: Oxaliplatin 130 mg/m2 IV on Day1, Capecitabine 825 or 1000 mg/m2 PO, BID Days on Days 1-14, Pembrolizumab 200 mg IV on Day 1.
  Safety validation: all Cycles are 21 days in length. Dose expansion: Cycle 1 is 28 days. Cycle 2 and beyond are 21 days.
Period: Overall Study
Arm/Group | Oxaliplatin + Capecitabine + Pembrolizumab
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The safety run-in was intended to identify dose-limiting toxicity. No DLTs were observed in the safety run-in and the drug dose levels were not changed in the expansion cohort, therefore; results were for safety validation and expansion were combined.
Groups:
- Oxaliplatin + Capecitabine + Pembrolizumab: For each cycle: Oxaliplatin 130 mg/m2 IV on Day1, Capecitabine 825 or 1000 mg/m2 PO, BID Days on Days 1-14, Pembrolizumab 200 mg IV on Day 1.
  Safety validation: all Cycles are 21 days in length. Dose Expansion: Cycle 1 is 28 days in length. Cycle 2 and beyond are 21 days.
Arm/Group | Oxaliplatin + Capecitabine + Pembrolizumab
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Months of Progression-free Survival (PFS)
Description: PFS measured from study entry until documented progression or death from any cause. Progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression. Patients who have not experienced progression will be censored at the date of the last radiographic assessment. The median PFS will be estimated using the Kaplan-Meier method.
Time Frame: Up to 44 months
Population: The safety run-in was intended to identify dose-limiting toxicity. No DLTs were observed in the safety run-in and the drug dose levels were not changed in the expansion cohort, therefore; results were for safety validation and expansion were combined. One treated patient did not complete cycle 1 of therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Oxaliplatin + Capecitabine + Pembrolizumab
Number analyzed (Participants) | 35
months | 7.6 [5.8 to 11.2]
Statistical Analysis 1: Comparison: Oxaliplatin + Capecitabine + Pembrolizumab; Test type: Superiority — 1-sided test of single exponential mean with historical null hypothesis of 5.5 months median PFS; p = 0.02, 1-sided exponential test — Sample size of 35 patients was chosen based on detecting the difference between a historical median PFS of 5.5 months and experimental median of 7.3 months, a hazard ratio of 0.75, with 80% power (1-sided test of single exponential mean, α=0.2)

2. Secondary Outcome: Response Rate as Measured by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: Response rate is calculated as the number of people with a complete response or partial response, divided by the total number of people treated. Complete response is defined as disappearance of all target lesions. Partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 44 months
Population: Treated patients with at least 1 re-staging. The safety run-in was intended to identify dose-limiting toxicity. No DLTs were observed in the safety run-in and the drug dose levels were not changed in the expansion cohort, therefore; results were for safety validation and expansion were combined.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Oxaliplatin + Capecitabine + Pembrolizumab
Number analyzed (Participants) | 33
proportion of participants | 0.76 [0. to 0.90]

3. Secondary Outcome: Months of Overall Survival
Description: Overall survival is the amount of time subjects live since starting the study.
Time Frame: Up to 44 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Oxaliplatin + Capecitabine + Pembrolizumab
Number analyzed (Participants) | 36
months | 16 [11.6 to 24.3]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug through 30 days after the last dose of study drug (up to 44 months).
Description: All grade 2-5 adverse events will be recorded in the study database. The safety run-in was intended to identify dose-limiting toxicity. No DLTs were observed in the safety run-in and the drug dose levels were not changed in the expansion cohort, therefore; results were for safety validation and expansion were combined.
Arm/Group | Oxaliplatin + Capecitabine + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 26/36
Serious Adverse Events (participants affected / at risk) | 17/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxaliplatin + Capecitabine + Pembrolizumab (N=36)
Pericardial tamponade (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 5
Colonic obstruction (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Sudden death NOS (General disorders) | 1
Device related infection (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Infections and infestations - Other, Specify (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic event (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxaliplatin + Capecitabine + Pembrolizumab (N=36)
Anemia (Blood and lymphatic system disorders) | 14
Sinus tachycardia (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 2
Endocrine disorders - Other, Specify (Endocrine disorders) | 1 — hypophysitis
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 3
Ascites (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 4
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 13
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 5
Esophageal pain (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 2
Fecal incontinence (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other, Specify (Gastrointestinal disorders) | 1 — anal itching
Gastrointestinal disorders - Other, Specify (Gastrointestinal disorders) | 1 — Abd cramping
Mucositis oral (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 15
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 10
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 14
Fever (General disorders) | 1
Gait disturbance (General disorders) | 1
Localized edema (General disorders) | 1
Malaise (General disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 2
Hepatobiliary disorders - Other, Specify (Hepatobiliary disorders) | 1 — hepatitis
Allergic reaction (Immune system disorders) | 1
Esophageal infection (Infections and infestations) | 1
Eye infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 2
Otitis externa (Infections and infestations) | 1
Otitis media (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 4
Wound infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Venous injury (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 5
Creatinine increased (Investigations) | 1
INR increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 11
Platelet count decreased (Investigations) | 3
Weight gain (Investigations) | 2
Weight loss (Investigations) | 9
White blood cell decreased (Investigations) | 9
Anorexia (Metabolism and nutrition disorders) | 15
Dehydration (Metabolism and nutrition disorders) | 7
Hyperglycemia (Metabolism and nutrition disorders) | 7
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 11
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 6
Hyponatremia (Metabolism and nutrition disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other, Specify (Metabolism and nutrition disorders) | 1 — failure to thrive/malnutrition
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, Specify (Musculoskeletal and connective tissue disorders) | 1 — R ankle
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Dysesthesia (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 3
Paresthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 13
Presyncope (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 5
Cystitis noninfective (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Nail loss (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 11
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Skin and subcutaneous tissue disorders - Other, Specify (Skin and subcutaneous tissue disorders) | 1 — rash at ankle, scalp, arms, left leg, nail changes
Skin and subcutaneous tissue disorders - Other, Specify (Skin and subcutaneous tissue disorders) | 1 — stage 2 skin breakdown to coccyx
Skin and subcutaneous tissue disorders - Other, Specify (Skin and subcutaneous tissue disorders) | 1 — scrotal rash, yeast
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 6
Hypotension (Vascular disorders) | 2
Superficial thrombophlebitis (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT03342937/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-09): https://cdn.clinicaltrials.gov/large-docs/37/NCT03342937/ICF_001.pdf